CLINICAL TRIAL: NCT06259110
Title: Revolutionizing Community-Acquired Pneumonia Diagnosis Through Integrating Novel Microbiological Techniques for Enhanced Precision
Brief Title: Community-Acquired Pneumonia Diagnosis Through Integrating Novel Microbiological Techniques.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Areej Osama Ali Mohammed Saleh, Assistant lecturer, Assiut University
Other Study IDs: CAP microbiological diagnosis
Record Dates: First submitted 2024-01-22; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Community-acquired Pneumonia
Keywords: Microbiological techniques; Multiplex PCR; Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multiplex PCR — multiplex PCR is a molecular biology technique that detect multiple respiratory pathogens including both bacteria and viruses from a single respiratory tract sample

SUMMARY:
To evaluate novel microbiological techniques for enhanced Pathogen Identification, assess the speed and efficiency of the integrated approach in providing timely diagnostic results, aiming to reduce the turnaround time for CAP diagnosis and subsequently improve patient outcomes and evaluate the clinical impact of enhanced precision in CAP diagnosis on treatment decisions, including the potential for targeted and more effective antimicrobial therapy based on accurate pathogen identification.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is the term used to describe an acute infection of the lungs that develops outside the hospital setting in a patient who has not been recently hospitalized.

Community-acquired pneumonia (CAP) is one of the most common infectious diseases and is a significant cause of mortality and morbidity globally despite preventative measures aimed at combating CAP.

These measures include pneumococcal vaccination of at-risk groups, yearly vaccinations for seasonal influenza viruses and since 2021, SARS-CoV-2 vaccination.

Understanding the etiology of CAP is crucial for accurate empirical antibiotic treatment, updating treatment guidelines, and future vaccine cost-benefit analyses. Currently, microbiological testing for CAP patients does not identify the etiology of most cases.

In contrast, molecular biology techniques, are rapid and sensitive for the diagnosis of pathogens. Furthermore, a multitude of nascent technologies, including multiplex real-time PCR; that detect multiple respiratory pathogens including both bacteria and viruses from a single respiratory tract sample and microarray methodologies, have become accessible for employment in clinical settings.

Improved diagnostics may change the management of CAP infections ,prompt identification of the appropriate organism would allow antibiotic de-escalation, which would decrease cost, adverse drug effects and antibiotic resistance pressure. These clinical interventions potentially translate to a reduced length of stay and financial savings for the patient, as well as an improved therapeutic outcome.

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinical diagnosis of pneumonia among both sexes
* Age >18 years Old.

Exclusion Criteria:

* Age <18 years old.
* Patients who refuse to participate in the study.
* patient who acquire infection after hospital admission within 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of pneumonia who acquire infection outside hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
. Evaluation of Novel Microbiological Techniques | baseline
  Measure sensitivity and specificity of novel microbiological techniques, such as rapid molecular tests, in identifying pathogens associated with CAP.

REFERENCES:
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Koo SH, Jiang B, Lim PQ, La MV, Tan TY. Development of a rapid multiplex PCR assay for the detection of common pathogens associated with community-acquired pneumonia. Trans R Soc Trop Med Hyg. 2021 Dec 2;115(12):1450-1455. doi: 10.1093/trstmh/trab079. PMID 34017992
- [Background] Naucler P, Henriques-Normark B, Hedlund J, Galanis I, Granath F, Ortqvist A. The changing epidemiology of community-acquired pneumonia: nationwide register-based study in Sweden. J Intern Med. 2019 Dec;286(6):689-701. doi: 10.1111/joim.12956. Epub 2019 Aug 13. PMID 31278792
- [Background] Demars Y, Brahier T, Rotzinger DC, Brouillet R, Jaton K, Opota O, Boillat-Blanco N. Utility of Polymerase Chain Reaction in Nasopharyngeal Swabs for Identifying Respiratory Bacteria Causing Community-Acquired Pneumonia. Microbiol Spectr. 2022 Jun 29;10(3):e0037922. doi: 10.1128/spectrum.00379-22. Epub 2022 May 18. PMID 35583335
- [Background] Nik Zuraina NMN, Mohamad S, Hasan H, Goni MD, Suraiya S. Diagnostic performance of an in-house multiplex PCR assay and the retrospective surveillance of bacterial respiratory pathogens at a teaching hospital, Kelantan, Malaysia. Pathog Glob Health. 2023 Feb;117(1):63-75. doi: 10.1080/20477724.2022.2028378. Epub 2022 Mar 25. PMID 35331083
- [Background] Hu L, Zhang S, Song W, Dong F, Xie Z, Chen X, Liu M, Cui B, Zhang Y, Zhang R, Wang Q. A sensitive mass spectrometry-based method to identify common respiratory pathogens in children. Microbiol Spectr. 2023 Sep 27;11(5):e0185823. doi: 10.1128/spectrum.01858-23. Online ahead of print. PMID 37754782
- See also: Dilemma-of-community-acquired-pneumonia — https://www.semanticscholar.org/paper/Dilemma-of-community-acquired-pneumonia-Shaaban/b7a7804c5b1e8e433dd23542d5ac32b7a63f9987